CLINICAL TRIAL: NCT00766207
Title: Preconception Risk Evaluation Via Electronic Medical Record Notification of Teratogenic Risks
Brief Title: Electronic Notification of Teratogenic Risks
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Eleanor Bimla Schwarz, MD, MS, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R18HS017093-01 (AHRQ); 1R18HS017093-01 (AHRQ)
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Teratogens; Abnormalities, Drug-Induced; Contraception
Keywords: Teratogens; Abnormalities, Drug-Induced; Contraception
MeSH Terms: conditions — Abnormalities, Drug-Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multi-faceted decision support (Experimental): Multi-faceted decision support
  Interventions: Other: Clinical decision support
- control (Active Comparator): stream-lined clinical alert
  Interventions: Other: stream-lined clinical alert

INTERVENTIONS:
Other: Clinical decision support — multi-faceted decision support
  Arms: multi-faceted decision support
Other: stream-lined clinical alert — electronic notification that a medication is potentially teratogenic
  Arms: control

SUMMARY:
This study will use a factorial design randomized controlled trial to (1)compare multi-faceted decision support (intervention) to streamlined clinical alerts (control) and (2) evaluate whether collecting information about women's risk of pregnancy using a networked tablet computer (intervention) is superior to the way clinicians usually collect this information (control).

Over the course of 1 year, we will abstract data from the electronic medical record when study clinicians prescribe teratogenic medications, conduct phone interviews with women prescribed medications by participating clinicians, and survey participating clinicians about their satisfaction with the decision support they receive. We will use this data to confirm our hypotheses that clinicians in the intervention groups will (1) prescribe fewer teratogenic medications, (2) be more likely to prescribe contraception when a teratogenic medication is prescribed, (3) have more patients report satisfaction with the counseling they received, and (4) report more satisfaction with the decision support they received.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 seen at a participating primary care clinic

Exclusion Criteria:

* Non-English speakers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2593 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Proportion of women prescribed potentially teratogenic medications with documented use of contraception | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor B Schwarz, MD, MS, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Partners in Health, Delmont, Pennsylvania
  - Partners in Health, Level Green, Pennsylvania
  - Partners in Health, Murrysville, Pennsylvania
  - General Internal Medicine Oakland (GIMO) Practice, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Schwarz EB, Parisi SM, Handler SM, Koren G, Cohen ED, Shevchik GJ, Fischer GS. Clinical decision support to promote safe prescribing to women of reproductive age: a cluster-randomized trial. J Gen Intern Med. 2012 Jul;27(7):831-8. doi: 10.1007/s11606-012-1991-y. PMID 22297687